CLINICAL TRIAL: NCT00115271
Title: Maternal Micronutrient Supplementation to Reduce Low Birth Weight and Infant and Maternal Morbidity in Rural Nepal
Brief Title: Antenatal Micronutrient Supplementation and Birth Weight
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency); Bill and Melinda Gates Foundation (Other); Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Parul Christian, Professor, Johns Hopkins Bloomberg School of Public Health
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: H.22.98.09.02.C1
Record Dates: First submitted 2005-06-21; First posted 2005-06-22 (Estimated); Last update posted 2014-08-26 (Estimated); Status verified 2014-08

CONDITIONS: Low Birth Weight; Infant Mortality; Pregnancy; Nutritional Status
Keywords: Micronutrients; Supplementation; Pregnancy; Birth weight; Infant mortality
MeSH Terms: conditions — Infant Death; Birth Weight | interventions — Dietary Supplements

INTERVENTIONS:
Drug: Nutritional supplements

SUMMARY:
The purpose of this study was to determine the effects of providing supplements containing alternative combinations of micronutrients during pregnancy on birth weight and other infant and maternal health and nutritional outcomes in a rural area of Nepal.

DETAILED DESCRIPTION:
Maternal micronutrient deficiencies are common in the developing world and may influence intrauterine growth and fetal and neonatal health and survival. Currently, policies for antenatal supplementation beyond iron-folic acid are not in place in these settings. And yet, the efficacy of such supplementation strategies has not been well established. Specifically, it is not clear if multiple micronutrient combinations will enhance fetal growth and newborn health and survival compared to single or smaller combinations of micronutrients. Also, while birth weight may serve as a proxy measure of newborn health, infant morbidity and mortality needs direct examination.

Comparisons: Pregnant women received daily folic acid, folic acid plus iron, folic acid plus iron plus zinc, or a multiple micronutrient supplement containing 11 other nutrients all with vitamin A compared to a control group that received only vitamin A.

ELIGIBILITY:
Inclusion Criteria:

* Married women of reproductive age identified as a new pregnancy using a urine test

Exclusion Criteria:

* Menopausal or sterilized woman or currently already pregnant or breastfeeding an infant <9 months of age

Ages: 15 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 5000
Dates: Start 1999-01; Primary Completion 2001-05 (Actual); Study Completion 2001-05 (Actual)

PRIMARY OUTCOMES:
Birth weight
3-month infant mortality

SECONDARY OUTCOMES:
Infant morbidity
Maternal morbidity
Maternal nutritional status
Weight gain during pregnancy
Infant growth

CONTACTS AND LOCATIONS:
Overall Officials: Parul Christian, DrPH, Principal Investigator — Johns Hopkins Bloomberg School of Public Health, Baltimore, MD 21205

REFERENCES:
- [Derived] Subedi S, Katz J, Erchick DJ, Verhulst A, Khatry SK, Mullany LC, Tielsch JM, LeClerq SC, Christian P, West KP, Guillot M. Does higher early neonatal mortality in boys reverse over the neonatal period? A pooled analysis from three trials of Nepal. BMJ Open. 2022 May 19;12(5):e056112. doi: 10.1136/bmjopen-2021-056112. PMID 35589346
- [Derived] Eroglu A, Schulze KJ, Yager J, Cole RN, Christian P, Nonyane BAS, Lee SE, Wu LSF, Khatry S, Groopman J, West KP Jr. Plasma proteins associated with circulating carotenoids in Nepalese school-aged children. Arch Biochem Biophys. 2018 May 15;646:153-160. doi: 10.1016/j.abb.2018.03.025. Epub 2018 Mar 30. PMID 29605494
- [Derived] Lee SE, Stewart CP, Schulze KJ, Cole RN, Wu LS, Yager JD, Groopman JD, Khatry SK, Adhikari RK, Christian P, West KP Jr. The Plasma Proteome Is Associated with Anthropometric Status of Undernourished Nepalese School-Aged Children. J Nutr. 2017 Mar;147(3):304-313. doi: 10.3945/jn.116.243014. Epub 2017 Feb 1. PMID 28148680
- [Derived] West KP Jr, Cole RN, Shrestha S, Schulze KJ, Lee SE, Betz J, Nonyane BA, Wu LS, Yager JD, Groopman JD, Christian P. A Plasma alpha-Tocopherome Can Be Identified from Proteins Associated with Vitamin E Status in School-Aged Children of Nepal. J Nutr. 2015 Dec;145(12):2646-56. doi: 10.3945/jn.115.210682. Epub 2015 Oct 7. PMID 26446483
- [Derived] Cole RN, Ruczinski I, Schulze K, Christian P, Herbrich S, Wu L, Devine LR, O'Meally RN, Shrestha S, Boronina TN, Yager JD, Groopman J, West KP Jr. The plasma proteome identifies expected and novel proteins correlated with micronutrient status in undernourished Nepalese children. J Nutr. 2013 Oct;143(10):1540-8. doi: 10.3945/jn.113.175018. Epub 2013 Aug 21. PMID 23966331
- [Derived] Christian P, Morgan ME, Murray-Kolb L, LeClerq SC, Khatry SK, Schaefer B, Cole PM, Katz J, Tielsch JM. Preschool iron-folic acid and zinc supplementation in children exposed to iron-folic acid in utero confers no added cognitive benefit in early school-age. J Nutr. 2011 Nov;141(11):2042-8. doi: 10.3945/jn.111.146480. Epub 2011 Sep 28. PMID 21956955
- [Derived] Christian P, Murray-Kolb LE, Khatry SK, Katz J, Schaefer BA, Cole PM, Leclerq SC, Tielsch JM. Prenatal micronutrient supplementation and intellectual and motor function in early school-aged children in Nepal. JAMA. 2010 Dec 22;304(24):2716-23. doi: 10.1001/jama.2010.1861. PMID 21177506
- [Derived] Lee AC, Darmstadt GL, Khatry SK, LeClerq SC, Shrestha SR, Christian P. Maternal-fetal disproportion and birth asphyxia in rural Sarlahi, Nepal. Arch Pediatr Adolesc Med. 2009 Jul;163(7):616-23. doi: 10.1001/archpediatrics.2009.75. PMID 19581544
- [Derived] Christian P, Darmstadt GL, Wu L, Khatry SK, Leclerq SC, Katz J, West KP Jr, Adhikari RK. The effect of maternal micronutrient supplementation on early neonatal morbidity in rural Nepal: a randomised, controlled, community trial. Arch Dis Child. 2008 Aug;93(8):660-4. doi: 10.1136/adc.2006.114009. PMID 18644934